CLINICAL TRIAL: NCT03070548
Title: A Phase 1 Open-label Study Of 14c-labeled Talazoparib In Patients With Advanced Solid Tumors
Brief Title: A Study of Talazoparib in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Medivation, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MDV3800-03; C3441003 (Other: Alias Study Number); 2016-001394-33 (EudraCT Number)
Record Dates: First submitted 2017-01-24; First posted 2017-03-03 (Actual); Results first posted 2018-12-17 (Actual); Last update posted 2018-12-17 (Actual); Status verified 2018-05

CONDITIONS: Advanced Solid Tumors
MeSH Terms: interventions — talazoparib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ADME (Experimental): 1 mg talazoparib containing100 μCi of 14C-radiolabeled talazoparib
  Interventions: Drug: Talazoparib

INTERVENTIONS:
Drug: Talazoparib — 1 mg of talazoparib containing100 μCi of 14C-radiolabeled talazoparib
  Other Names: MDV3800; BMN673

SUMMARY:
This study will evaluate the mass balance of talazoparib after a single dose of talazoparib.

DETAILED DESCRIPTION:
Patients participating in this study with no clinically significant toxicities may be eligible to continue treatment on a separate extension protocol after discussion with the Principal Investigator and obtaining Sponsor permission..

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age and willing and able to provide informed consent.
2. Histologically confirmed advanced solid tumor (limited to platinum-resistant ovarian carcinoma, cervical adenocarcinoma, small cell lung carcinoma or triple-negative breast cancer) judged by the Investigator to not be appropriate for standard therapy.
3. Eastern Co-Operative Oncology Group (ECOG) performance status ≤ 2 at screening and Day -1.
4. Expected life expectancy of ≥ 3 months.
5. Able to swallow the study drug and comply with study requirements.
6. Female subjects may be enrolled if they are considered not of childbearing potential, or who are post-menopausal, or of childbearing potential using a highly effective form of contraception, and female subjects should not donate eggs from the time point of IMP administration until at least 45 days thereafter.
7. Males with partners of childbearing potential may be enrolled if they use a condom when having sex with a pregnant woman or with a woman of childbearing potential from 21 days before the first dose of study drug through 105 days after the last dose of study drug, and males should not donate sperm from the time point of study drug administration until at least 105 days thereafter.
8. Female patients must not be breastfeeding at screening and during the study participation until 45 days after the last dose of the study drug.
9. Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests, and other trial procedures.

Exclusion Criteria:

1. Treatment within 14 weeks or five half-live prior to dosing with any type of systemic anticancer therapy or any investigational agent, whichever is longer.
2. Major surgery within 8 weeks before screening.
3. Serious accompanying disorder or impaired organ function.
4. Symptomatic or impending spinal cord compression or cauda equina syndrome.
5. Non-healing wound, ulcer, or bone fracture, not including a pathological bone fracture caused by a pre-existent pathological bone lesion.
6. Known myelodysplastic syndrome.
7. Patients with the following serologies should be excluded: HBsAg+ or anti-HBc+; HCV+; HIV+.
8. Serious or unstable medical condition that interferes with ability to tolerate treatment or assessments associated with the protocol.
9. Gastrointestinal disorder affecting absorption.
10. Known hypersensitivity to any of the talazoparib solution components.
11. Use of a strong P-gp inhibitor, strong P-gp inducer, or strong inhibitor of BRCP within 7 days or 5 half-lives, whichever is longer, before Day 1.
12. Any condition or reason that interferes with ability to participate in the study, causes undue risk, or complicates the interpretation of safety data, in the opinion of the Investigator or Sponsor (e.g. non-compliance, excessive alcohol consumption, intake of drugs of abuse unless these drugs are medically indicated [e.g. opiates for pain relief]).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2016-09 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- PRA Magyarorszag Kft, Fazis I-es Klinikai Farmakologiai Vizsgalohely, Budapest, Hungary

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=MDV3800-03&StudyName=A+Phase+1+Open-label%2C+Two-arm%2Cdrug-drug+Interaction+Study+To+Evaluate+The+Effect+Of+Itraconazole+And+Rifampin+On+The+Pharmacokinetics+Of+Talazoparib+In+Patients+With+Advanced+Solid+Tumors
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=MDV3800-03&StudyName=A+Phase+1+Open-label+Study+Of+14c-labeled+Talazoparib+In+Patients+With+Advanced+Solid+Tumors

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This is a mass balance study with 14C-radiolabeled talazoparib in at least 6 participants with advanced solid tumors who qualified for treatment with talazoparib. Participants who completed the mass-balance part in this study had the option to continue treatment on an open-label extension protocol.
Groups:
- Talazoparib: Participants with advanced solid tumors received a single dose of talazoparib 1 miligram (mg) oral solution (containing approximately 100 micro Curie of 14C-talazoparib) on Day 1. Participants were followed-up within 14 days after the last day of mass balance phase and at least 30 days after Day 1 or the first day of extension protocol, whichever occurred first (up to maximum duration of 8 weeks from screening to follow-up for each participant).
Period: Overall Study
Arm/Group | Talazoparib
Started | 6
Completed | 6
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Safety analysis set included all participants who had received at least 1 dose of study drug.
Groups:
- Talazoparib: Participants with advanced solid tumors received a single dose of talazoparib 1 mg oral solution (containing approximately 100 micro Curie of 14C-talazoparib) on Day 1. Participants were followed-up within 14 days after the last day of mass balance phase and at least 30 days after Day 1 or the first day of extension protocol, whichever occurred first (up to maximum duration of 8 weeks from screening to follow-up for each participant).
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
Age, Continuous [Mean (Standard Deviation); unit: years] | 50.2 (17.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 6
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 6
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of Talazoparib
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: Pharmacokinetic (PK) population included all participants who received talazoparib and had at least 1 sample with sufficient concentration data.
Measure: Mean (Standard Deviation); unit: nanogram per milliliter (ng/mL)
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
nanogram per milliliter (ng/mL) | 8.4 (3.8)

2. Primary Outcome: Time to Attain Maximum Observed Plasma Concentration (Tmax) of Talazoparib
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: PK population included all participants who received talazoparib and had at least 1 sample with sufficient concentration data.
Measure: Median (Full Range); unit: hours
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
hours | 0.5 [0.5 to 0.5]

3. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of Talazoparib
Description: AUC(0-inf) was defined as the area under the plasma concentration-time curve from time zero (pre-dose) to extrapolated infinite time (0-inf).
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram per milliliter (hr*ng/mL)
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
hour*nanogram per milliliter (hr*ng/mL) | 129.9 (70.4)

4. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC0-last) of Talazoparib
Description: AUC(0-last) was defined as the area under the plasma concentration-time curve from zero to the time of the last measurable concentration.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hr*ng/mL
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
hr*ng/mL | 118.9 (65.4)

5. Primary Outcome: Terminal Elimination Half-Life (t1/2) of Talazoparib
Description: Terminal elimination half-life was defined as time measured for the plasma concentration of talazoparib to decrease by one half.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
hours | 89.8 (57.6)

6. Primary Outcome: Apparent Total Plasma Clearance (CL/F) of Talazoparib
Description: Clearance of a drug was measure of the rate at which a drug was metabolized or eliminated by normal biological processes.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
liter/hour | 8.39 (3.7)

7. Primary Outcome: Apparent Volume of Distribution (Vd/F) of Talazoparib
Description: Apparent volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of the drug.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
liter | 922.6 (445.8)

8. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) of 14C- Radioactivity
Description: 100 micro-curie of 14C-radiolabeled talazoparib was present in 1 mg of talazoparib.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram equivalent/mililiter
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
nanogram equivalent/mililiter | 12.1 (5.8)

9. Primary Outcome: Time to Attain Maximum Observed Plasma Concentration (Tmax) of 14C- Radioactivity
Description: 100 micro-curie of 14C-radiolabeled talazoparib was present in 1 mg of talazoparib.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
hours | 0.5 [0.5 to 0.5]

10. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of 14C- Radioactivity
Description: AUC(0-inf) was defined as the area under the plasma concentration-time curve from time zero (pre-dose) to extrapolated infinite time (0-inf). 100 micro-curie of 14C-radiolabeled talazoparib was present in 1 mg of talazoparib.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram equivalent/mililiter
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
hour*nanogram equivalent/mililiter | 222.9 (108.8)

11. Primary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC0-last) of 14C- Radioactivity
Description: AUC(0-last) was defined as the area under the plasma concentration-time curve from zero to the time of the last measurable concentration. 100 micro-curie of 14C-radiolabeled talazoparib was present in 1 mg of talazoparib.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram equivalent/mililiter
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
hour*nanogram equivalent/mililiter | 199.3 (101.9)

12. Primary Outcome: Terminal Elimination Half-Life (t1/2) of 14C- Radioactivity in Plasma
Description: Terminal elimination half-life was defined as the time measured for the plasma radioactivity concentration to decrease by one half. 100 micro-curie of 14C-radiolabeled talazoparib was present in 1 mg of talazoparib.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
hours | 96.2 (55.1)

13. Primary Outcome: Apparent Total Plasma Clearance (CL/F) of 14C- Radioactivity
Description: Clearance of a drug was a measure of the rate at which a drug was metabolized or eliminated by normal biological processes. 100 micro-curie of 14C-radiolabeled talazoparib was present in 1 mg of talazoparib.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
liter/hour | 5.35 (2.35)

14. Primary Outcome: Apparent Volume of Distribution (Vd/F) of 14C- Radioactivity in Plasma
Description: Apparent volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of a drug. 100 micro-curie of 14C-radiolabeled talazoparib was present in 1 mg of talazoparib.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
liter | 655.8 (338.1)

15. Primary Outcome: Maximum Observed Whole Blood Concentration (Cmax) of 14C- Radioactivity
Description: 100 micro-curie of 14C-radiolabeled talazoparib was present in 1 mg of talazoparib.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: nanogram equivalent/mililiter
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
nanogram equivalent/mililiter | 12.5 (5.7)

16. Primary Outcome: Time to Attain Maximum Observed Whole Blood Concentration (Tmax) of 14C- Radioactivity
Description: 100 micro-curie of 14C-radiolabeled talazoparib was present in 1 mg of talazoparib.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
hours | 0.5 [0.5 to 0.5]

17. Primary Outcome: Area Under the Whole Blood Concentration-Time Curve From Time Zero to Infinity (AUC0-inf) of 14C- Radioactivity
Description: as for outcome 10
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram equivalent/mililiter
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
hour*nanogram equivalent/mililiter | 234.1 (114.1)

18. Primary Outcome: Area Under the Whole Blood Concentration-Time Curve From Time Zero to Last Quantifiable Concentration (AUC0-last) of 14C- Radioactivity
Description: as for outcome 11
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: hour*nanogram equivalent/mililiter
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
hour*nanogram equivalent/mililiter | 205.8 (101.0)

19. Primary Outcome: Apparent Total Whole Blood Clearance (CL/F) of 14C- Radioactivity
Description: as for outcome 13
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
liter/hour | 5.21 (2.51)

20. Primary Outcome: Apparent Volume of Distribution (Vd/F) of 14C- Radioactivity in Whole Blood
Description: Apparent volume of distribution was defined as the theoretical volume in which the total amount of drug would need to be uniformly distributed to produce the desired plasma concentration of the drug. 100 micro-curie of 14C-radiolabeled talazoparib was present in 1 mg of talazoparib.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
liter | 484.4 (237.5)

21. Primary Outcome: Amount of Talazoparib Excreted in Urine During Each Collection Interval (Ae t1-t2)
Description: Ae t1-t2 was defined as the amount of talazoparib excreted into urine during each collection interval (t1-t2).
Time Frame: Pre-dose, 0 to 8 hours (hrs), 8 to 24 hrs, 24 to 48 hrs, 48 to 72 hrs, 72 to 96 hrs and then after every 24 hrs until up to 504 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: micrograms
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
micrograms | 366.07 (45.56)

22. Primary Outcome: Percentage of Dose of Talazoparib Excreted During Each Collection Interval (Aet1-t2%) of Talazoparib
Description: Aet1-t2% was the percentage of Aet1-t2, where Aet1-t2 was defined as the amount of talazoparib excreted into urine during each collection interval (t1-t2).
Time Frame: Pre-dose, 0 to 8 hrs, 8 to 24 hrs, 24 to 48 hrs, 48 to 72 hrs, 72 to 96 hrs and then after every 24 hrs until up to 504 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
percentage of dose | 40.92 (4.324)

23. Primary Outcome: Renal Clearance (CLr) of Talazoparib
Description: Renal clearance was calculated as cumulative amount of drug excreted in urine divided by AUC(0-last) (area under the plasma concentration-time curve from zero to the time of the last measurable concentration).
Time Frame: as for outcome 22
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: liter/hour
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
liter/hour | 3.808 (1.979)

24. Primary Outcome: The Recovery of 14C-Radioactivity as a Percentage of the Administered Dose
Description: Recovery of 14C-radioactivity in urine and feces was calculated in terms of percentage of administered dose after administration of a single 1 mg dose of oral solution (containing 100 micro-curie 14C-labeled talazoparib).
Time Frame: From 0 to 8 hrs, 8 to 24 hrs, 24 to 48 hrs and then after every 24 hrs until up to 504 hrs post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percentage of dose
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
Percentage of dose
  Urine | 68.647 (8.592)
  Feces | 19.669 (5.493)

25. Secondary Outcome: Ratio of Maximum Observed Plasma Concentration to Maximum Observed Whole Blood Concentration for 14C- Radioactivity
Description: 100 micro-curie of 14C radiolabeled talazoparib was present in 1 mg of talazoparib.
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
ratio | 1.050 (0.0625)

26. Secondary Outcome: Ratio of Area Under the Plasma Concentration-Time Curve From Time Zero to Infinity to Area Under the Whole Blood Concentration-Time Curve From Time Zero to Infinity for 14C- Radioactivity
Description: as for outcome 10
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
ratio | 1.047 (0.1155)

27. Secondary Outcome: Ratio of Area Under the Plasma Concentration-Time Curve From Time Zero to Last Quantifiable Concentration to Area Under the Whole Blood Concentration-Time Curve From Time Zero to Last Quantifiable for 14C- Radioactivity
Description: as for outcome 11
Time Frame: Pre-dose, 0.5, 1, 2, 4, 8, 12, 24, 48, 72, 96, 120, 168, 216, 264, 336, 384, 432 and 504 hours post-dose
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
ratio | 1.037 (0.1243)

28. Secondary Outcome: Number of Participants With Treatment Emergent Adverse Events (AEs)
Description: An AE was any untoward medical occurrence in a participant who received study drug without regard to possibility of causal relationship. Treatment-emergent were events between first dose of study drug through 14 days after the last day of mass balance phase and at least 30 days after Day 1 or before initiation of new cytotoxic chemotherapy, new investigational treatment, or the first day of extension protocol, whichever occurs first (up to maximum duration of 8 weeks from screening to follow-up for each participant) or before initiation of new cytotoxic chemotherapy, new investigational treatment, or the first day of extension protocol, whichever occurs first, that were absent before treatment or that worsened relative to pre-treatment state. AEs included both non-serious (AEs) and serious adverse events (SAEs).
Time Frame: Day 1 to 14 days after last day of mass balance phase and at least 30 days after Day1/before initiation of new cytotoxic chemotherapy, new investigational treatment/first day of extension protocol, whichever occurs first(up to maximum duration of 8 weeks)
Population: Safety analysis set included all participants who received at least 1 dose of talazoparib.
Measure: Number; unit: participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
participants | 4

29. Secondary Outcome: Number of Participants With Clinically Significant Vital Signs Parameters
Description: Vital Signs included heart rate, respiratory rate, body temperature, systolic blood pressure and diastolic blood pressure. clinical significance of vital signs was determined at the investigator's discretion.
Time Frame: Baseline up to Day 22
Population: Safety analysis set included all participants who received at least 1 dose of talazoparib.
Measure: Number; unit: participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
participants | 0

30. Secondary Outcome: Number of Participants With Clinically Significant Electrocardiogram (ECG) Abnormalities
Description: Criteria for clinically significant ECG abnormalities : Heart Rate; increase from baseline greater than (>)25 %and to a value >100, decrease from baseline >25% and to a value < 50; PR Interval: increase from baseline >25% and to a value >200; QRS Duration: increase from baseline >25% and to a value >100; QT interval using Fridericia's correction (QTcF): ranges >450 msec, >480 msec, >500 msec, Increase from baseline >30 msec and >60 msec; QT Interval: ranges >450 msec, >480 msec, >500 msec, Increase from baseline >30 msec and >60 msec.
Time Frame: Baseline up to Day 22
Population: Safety population set included all participants who received at least 1 dose of talazoparib.
Measure: Number; unit: participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
participants | 0

31. Secondary Outcome: Number of Participants With Clinically Significant Laboratory Abnormalities
Description: Haematological, biochemistry and urinalysis parameters. Biochemistry parameters:alkaline phosphatase 30-120units per liter(U/L), creatinine 53-110micromole/L(micromol/L), gamma glutamyl transferase 7-50U/L, glucose 3.3-5.5millimoles/L(mmol/L), lactate dehydrogenase 200-460U/L, triglycerides 0.4-1.7mmol/L, cholesterol 2.6-5.2mmol/L, phosphate 0.8-1.45mmol/L, sodium 135-146mmol/L, urea 2.8-7.2mmol/L, chloride 95-109mmol/L, creatine kinase 24-170U/L, aspartate aminotransferase 4-46U/L, potassium 3.5-5.5mmol/L. Haematology parameters:haemoglobin 120-155 gram/L(g/L), erythrocytes 4-5.2 10^12/L, haematocrit 0.35-0.45, prothrombin time 13.7-15.6 second(sec), lymphocytes 1-3.7 10^9/L, platelets 150-400 10^9/L, prothrombin intl. normalized ratio 0.89-1.1, activated partial thromboplastin time 25-43 sec, basophils 0-0.09 10^9/L, neutrophils 1.5-7 10^9/L, and leukocytes 4-10 10^9/L. Urinalysis parameters:urinalysis specific gravity 1.012-1.03, urinalysis pH 4.8-7.8.
Time Frame: Baseline up to Day 22
Population: Safety population set included all participants who received at least 1 dose of talazoparib.
Measure: Number; unit: participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
participants | 0

32. Secondary Outcome: Number of Participants With Change From Baseline in Physical Examination Findings
Description: Physical examination included examination of abdomen, cardiovascular, eyes, ears, nose, throat, general appearance, head, neck, thyroid, lymph nodes, musculoskeletal, neurological, skin/subcutaneous tissue and thorax/lungs.
Time Frame: Baseline up to Day 22
Population: Safety population set included all participants who received at least 1 dose of talazoparib.
Measure: Number; unit: participants
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
participants | 0

33. Secondary Outcome: Amount of Any Significant Metabolites of Talazoparib in Urine and Feces
Description: M4 (M481/1, cysteine conjugate of mono-desfluoro-talazoparib) metabolite was found in urine. MDV10595 (M1, dehydrogenated talazoparib (PF-07052386), M556/1 (glucuronide conjugate of talazoparib), and M2 (M396/1, mono-oxidative talazoparib) metabolites were calculated together and were also found in urine. Three metabolites named as: MDV10595 (M1)/M556/1 and M2 (M396/1) which were calculated together were detected in feces. Amount of metabolite in this outcome measure was measured in terms of percentage of dose of talazoparib.
Time Frame: From 0 to 8 hrs, 8 to 24 hrs, 24 to 48 hrs and then after every 24 hrs until up to 504 hrs post-dose
Population: as for outcome 2
Measure: Number; unit: percentage of dose
Arm/Group | Talazoparib
Number analyzed (Participants) | 6
percentage of dose
  M481/1: Urine | 4.2
  MDV10595+M556/1+M396/1: Urine | 0.8
  MDV10595+M556/1+M396/1: Feces | 1.5

ADVERSE EVENTS:
Time Frame: Day1 up to 14days after last day of mass balance phase and at least 30days after Day1/ before initiation of new cytotoxic chemotherapy, new investigational treatment/ first day of extension protocol, whichever occurs first (up to maximum duration of 8weeks from screening to follow-up for each participant)
Description: Same event may appear as AE and SAE, what is presented are distinct events. Event may be categorized as serious in 1 participant and as non-serious in another participant or 1 participant may have experienced both serious and non-serious event during study. Safety analysis set included all participants who had received at least 1 dose of study drug.
Arm/Group | Talazoparib
All-Cause Mortality (participants affected / at risk) | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6
Other Adverse Events (participants affected / at risk) | 4/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Talazoparib (N=6)
Constipation (Gastrointestinal disorders) | 1
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Dizziness (Nervous system disorders) | 2
Pollakiuria (Renal and urinary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2016-10-07): https://cdn.clinicaltrials.gov/large-docs/48/NCT03070548/Prot_000.pdf
  • Statistical Analysis Plan (2017-07-16): https://cdn.clinicaltrials.gov/large-docs/48/NCT03070548/SAP_001.pdf